CLINICAL TRIAL: NCT02218931
Title: Effect of Simple, Targeted Diet in Pregnant Women With Metabolic Risk Factors on Pregnancy Outcomes (ESTEEM): A Randomised Trial
Brief Title: ESTEEM - Effect of Simple, Targeted Diet in Pregnant Women With Metabolic Risk Factors on Pregnancy Outcomes
Acronym: ESTEEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 009337QM; 732/2029 (Other Grant/Funding Number: Barts Charity)
Record Dates: First submitted 2014-07-11; First posted 2014-08-18 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-01

CONDITIONS: Pre-eclampsia; Obesity; Raised Lipids; High Blood Pressure; Insulin Resistance; Gestational Diabetes; Small for Gestational Age; Stillbirth
Keywords: Pre-eclampsia; Gestational diabetes; Stillbirth; Small for gestational age; Admission to neonatal intensive care unit; Obesity; Raised Lipids; High Blood Pressure; Cardiovascular risk; Insulin resistance; Mediterranean dietary pattern; Dietary interventions
MeSH Terms: conditions — Pre-Eclampsia; Obesity; Hypertension; Insulin Resistance; Diabetes, Gestational; Stillbirth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Targeted ESTEEM diet (Experimental): The ESTEEM dietary pattern is similar to that in a Mediterranean diet associated with reduced risk of pre-eclampsia.
  The intervention will include structured meal plans and grocery lists, recipes for healthy diet and appropriate choices at restaurants
  Interventions: Behavioral: Targeted ESTEEM diet
- Current clinical practice (No Intervention): The control group will be provided the usual antenatal dietary advice. This includes advice on healthy and physical activity in women with normal weight and obesity and overweight. Folic acid and vit D supplementation are provided as per national recommendations. Participants will provide outcome data at point of delivery and food frequency questionnaire at baseline and 36 weeks or delivery depending on which is sooner.
- Non-randomised cohort (Other): Non-randomised cohort of women with no metabolic risk factors will be followed up to delivery to collect outcome data
  Interventions: Other: Non-randomised cohort

INTERVENTIONS:
Behavioral: Targeted ESTEEM diet — The key components of the diet are:
  High intake of vegetables, nuts, non-refined grains, legumes and fruits;Moderate to high consumption of fish;Small to moderate intake of poultry and dairy products such as yoghurt and cheese;Low consumption of red meat and processed meat and avoidance of sugary drinks, fast food and high fat food;High fibre;Intake of nuts including walnuts and almonds that are rich sources of monounsaturated and polyunsaturated fatty acids (30 g/day);Olive oil to cook and dress salads as the main source of fat (0.5 l/week)
  The intervention will include structured meal plans and grocery lists, recipes for healthy diet and appropriate choices at restaurants
  Arms: Targeted ESTEEM diet
Other: Non-randomised cohort — Non-randomised cohort of women with no metabolic risk factors will be followed up to delivery to collect outcome data
  Arms: Non-randomised cohort

SUMMARY:
Obesity is a growing problem in East London and every other woman who enters pregnancy is obese or overweight. In addition to obesity, other metabolic risk factors such as raised lipids, high blood pressure and diabetes increase pregnancy related complications such as preeclampsia and long term problems such as heart diseases, stroke and death. Preeclampsia, presenting as hypertension and proteinuria is a leading cause of maternal and fetal mortality and morbidity. Interventions that reduce cardiovascular events by modifying risk factors also have the potential to reduce the risk of preeclampsia. The investigators work funded by the National Institute of Health Research (NIHR) in the UK showed that dietary interventions in obese pregnant women may reduce the risk of preeclampsia. The investigators propose to show that pregnant women with metabolic risk factors derive the most benefit from a simple, targeted intervention based on Mediterranean dietary pattern to reduce the risk of maternal and fetal complications . Women with the risk factors (1230 women) will be randomly allocated to dietary intervention or usual antenatal dietary advice and the risk of maternal and fetal complications will be evaluated. The remaining eligible women who are consented for lipid tests, but do not have metabolic risk factors, will be followed up for outcome data only. Diet based interventions, especially those based on a Mediterranean dietary pattern has a potential to reduce the risk of preeclampsia. In the investigators study, pregnant mothers with risk factors will be randomly allocated to either a dietary invention or usual antenatal care and they will assess their composite maternal (pre-eclampsia or gestational diabetes) and fetal (stillbirth, small for gestational age or admission to neonatal intensive care unit) outcomes. The investigators will tailor the intervention to suit the individual needs of the mother and provide nuts and olive oil to improve compliance. The study will be undertaken across the three maternity units at Barts Health NHS Trust, which delivers 17,000 women/year and two other maternity units in England. The study is supported by the office of the Mayor of Tower Hamlets which will facilitate the involvement of grassroots workers to promote recruitment and uptake of the intervention.

DETAILED DESCRIPTION:
Obesity is a growing problem in east London with a fifth of women entering pregnancy as obese. In addition to obesity, other metabolic risk factors such as raised lipids, high blood pressure and insulin resistance are increasingly prevalent. With a large proportion of ethnic minority mothers in east London, dietary habits and underlying genetic predisposition are major contributors to this phenomenon. Obesity and raised serum lipids, especially triglycerides increase the risk of complications such as preeclampsia in pregnancy and cardiovascular events such as myocardial infarction, stroke and death in the long term. Preeclampsia, a condition in pregnancy, with raised blood pressure and increased protein in the urine is a leading cause of maternal and fetal deaths. Its treatment gives rise to large health care costs. Preeclampsia contributes to preterm birth, one of the leading causes of perinatal deaths in east London. It accounts for 65% of neonatal deaths and 50% of neurological disability in childhood. Around £900 million in extra costs for care of preterm babies per year in the NHS are linked to neonatal care. Preeclampsia, characterised by insulin resistance, widespread endothelial damage and dysfunction, coagulation defects and increased systemic inflammatory response, shares metabolic risk factors with cardiovascular disease. Obesity, dyslipidaemia and hypertension are independent risk factors for pre-eclampsia. Interventions that reduce cardiovascular events by modifying metabolic risk factors also have the potential to reduce the risk of pre-eclampsia.

Early identification of mothers at risk of preeclampsia will allow clinicians to deliver these targeted interventions in pregnancy, with the potential to prevent preeclampsia and modify cardiovascular risk in the long-term. Currently, low dose aspirin, recommended as a prophylactic measure reduces preeclampsia risk by only 10%. Simple, low-cost and effective acceptable interventions are required to reduce this risk further. Dietary interventions in pregnant women with metabolic risk factors such as obesity and insulin resistance are shown to reduce the risk of preeclampsia. But the existing studies are of poor quality and do not evaluate preeclampsia as the primary outcome. Furthermore, they focus on specific components of the diet, rather than modifying the overall dietary pattern. Mediterranean diet with high consumption of vegetables and fruits, olive oil and nuts and low consumption of red meat and processed food significantly reduces lipid levels and cardiovascular adverse events in non-pregnant high risk population. In pregnancy, the beneficial effect of the Mediterranean dietary pattern was observed in a large prospective study of nulliparous pregnant women with a 28% reduction in the risk of preeclampsia (RR 0.72; 95% CI 0.62, 0.85). These results need confirmation in a sound experimental study.

There is a need for an adequately powered randomised trial to evaluate the beneficial effect of lipid modifying diet in pregnancy that is simple, accessible and acceptable. The investigators hypothesis is that pregnant women with metabolic risk factors will derive benefit from dietary intervention in preventing maternal and fetal complications.

ELIGIBILITY:
Inclusion Criteria: Pregnant women less than 18 weeks of gestation with at least one of the following:

i. BMI ≥30 Kg/m2 ii. Raised serum triglycerides ≥1.7 mmol/l iii. Raised blood pressure of systole ≥140 mm Hg or diastole ≥90 mm Hg

Exclusion Criteria:

i. BMI <18.5 Kg/m2or ≥40 Kg/m2 ii. Women on lipid altering drugs iii. History of diabetes iv. Chronic renal disease v. Auto immune disease vi. Multiple pregnancy vii. Poor understanding of written and spoken English viii. Not able to follow Mediterranean diet for religious or other reasons ix. <16 years of age x. Not able to consume nuts or extra virgin olive oil

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3442 (Actual)
Dates: Start 2014-09-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Composite maternal outcomes: pre-eclampsia or gestational diabetes | At delivery
  Diagnosis of pre-eclampsia defined as:
  * new onset hypertension after 20 weeks gestation defined as systolic BP ≥ 140 mm Hg or diastolic BP ≥ 90 mmHg, in at least two readings AND New onset proteinuria defined as spot urine Protein/creatinine ratio (PCR) test greater than 30mg/mmol or >24 hour urine 300mg/24 hours or 2+ or more on standard urinary dipstick tests after 20 weeks gestation
  * superimposed pre-eclampsia in women with chronic hypertension or chronic proteinuria
  * women with eclamptic seizures with no hypertension or proteinuria
  Diagnosis of gestational diabetes defined as:
  * fasting venous glucose of 5·1 mmol/L or higher or
  * 2 h venous glucose of 8·5 mmol/L or higher or
  * combination of these
Composite fetal outcomes: stillbirth, small for gestational age or admission to neonatal intensive care unit | At delivery

SECONDARY OUTCOMES:
To assess the effect of targeted dietary intervention vs. usual antenatal dietary advice on other maternal and fetal outcomes | At delivery
The number of participants with a change in lipid profiles from early pregnancy to delivery in women a) with and without dietary interventions b) with and without pre-eclampsia on the composite maternal and fetal outcomes. | At delivery
The rates of composite maternal and fetal outcomes in the following subgroups of women in the intervention and control group: obese; raised triglycerides and with raised blood pressure. | Baseline and 36 weeks or delivery depending on which is sooner
Development of a cohort for medium and long term follow up of mothers and babies after birth through applications to other grant giving bodies. | End of follow up, an average of 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Shakila Thangaratinam, Principal Investigator — Queen Mary University of London; Rehan Khan, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] H Al Wattar B, Dodds J, Placzek A, Beresford L, Spyreli E, Moore A, Gonzalez Carreras FJ, Austin F, Murugesu N, Roseboom TJ, Bes-Rastrollo M, Hitman GA, Hooper R, Khan KS, Thangaratinam S; ESTEEM study group. Mediterranean-style diet in pregnant women with metabolic risk factors (ESTEEM): A pragmatic multicentre randomised trial. PLoS Med. 2019 Jul 23;16(7):e1002857. doi: 10.1371/journal.pmed.1002857. eCollection 2019 Jul. PMID 31335871
- [Derived] Al Wattar BH, Dodds J, Placzek A, Spyreli E, Higgins S, Moore A, Hooper R, Beresford L, Roseboom TJ, Bes-Rastrollo M, Hitman G, Khan KS, Thangaratinam S; ESTEEM study group. Mediterranean diet based intervention in pregnancy to improve maternal and fetal outcomes: Methodological challenges and lessons learned from the multicentre ESTEEM study. Contemp Clin Trials Commun. 2017 Mar 29;6:72-77. doi: 10.1016/j.conctc.2017.02.012. eCollection 2017 Jun. PMID 29740638
- [Derived] Al Wattar BH, Dodds J, Placzek A, Spyreli E, Moore A, Hooper R, Beresford L, Roseboom TJ, Bes-Rastrollo M, Hitman G, Khan KS, Thangaratinam S; ESTEEM study group. Effect of simple, targeted diet in pregnant women with metabolic risk factors on maternal and fetal outcomes (ESTEEM): study protocol for a pragmatic multicentre randomised trial. BMJ Open. 2016 Oct 21;6(10):e013495. doi: 10.1136/bmjopen-2016-013495. PMID 27798035